CLINICAL TRIAL: NCT01460862
Title: Analyze the Impact of Omalizumab on Corticosteroid Use, Emergency Room Visits and Hospitalizations Among Patients With Uncontrolled Asthma Receiving High Dose Inhaled Corticosteroids
Brief Title: Impact of Omalizumab on Corticosteroid Use, Emergency Room Visits and Hospitalizations
Status: Withdrawn | Type: Observational
Why Stopped: company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: HEORUS0091
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: Asthma; Omalizumab
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Omalizumab Cohort

SUMMARY:
A retrospective database analysis to evaluate the impact of omalizumab on the use of corticosteroid, emergency-department visits and hospitalizations among patients with uncontrolled asthma and using high-dose Inhaled Corticosteroids (ICS) prior to initiating omalizumab.

ELIGIBILITY:
Inclusion Criteria:

* ≥12 years of age with a documented Cystic fibrosis (CF) diagnosis,
* on Long acting Beta antagonist- Inhaled Corticosteroid (LABA-ICS) at baseline,
* uncontrolled asthma at baseline.

Exclusion Criteria:

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with uncontrolled asthma and using high-dose ICS prior to initiating omalizumab.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05 (Estimated); Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of emergency-department visits and hospitalizations | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals